CLINICAL TRIAL: NCT04915846
Title: TAM4MTM: a Phase 1/2 Randomized, Placebo-Controlled, Double-Blinded, Single Crossover Study to Determine the Safety and Efficacy of Tamoxifen Therapy for Myotubular Myopathy (XLMTM)
Brief Title: Tamoxifen Therapy for Myotubular Myopathy
Acronym: TAM4MTM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to safety concerns.
Sponsor: James Dowling (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Cures Within Reach (Other); The Joshua Frase Foundation USA (Unknown); Will Cure USA (Unknown); Mogford Campbell Family Chair Fund (Unknown); Myotubular Trust (Unknown); Great Ormond Street Hospital Charity (Unknown); Sparks (Unknown)
Responsible Party: Sponsor-Investigator, James Dowling, Staff clinician and senior scientist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAM4MTM / OZM-098
Record Dates: First submitted 2021-05-06; First posted 2021-06-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: X Linked Myotubular Myopathy
Keywords: tamoxifen; X-linked myotubular myopathy
MeSH Terms: conditions — Myopathies, Structural, Congenital | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-controlled, single cross-over study with washout period before cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is a placebo-controlled double-blinded design. A select few (pharmacist and study staff in charge of pharmacokinetics) and Data Safety Monitoring Board (DSMB) are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: ApoTamox 10mg (Experimental): Drug: Tamoxifen (tamoxifen citrate); ApoTamox 10 mg tablets orally twice daily for 6 months
  Interventions: Drug: ApoTamox 10mg
- Placebo (Placebo Comparator): Placebo (no active ingredients) tablets orally twice daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ApoTamox 10mg — All participants will receive tamoxifen (ApoTamox) for approximately 6 months (6 months + 1 week). Participants and study staff will be blinded as to whether the participants are starting with the placebo or the drug. Depending on randomization, drug or placebo will be dispensed at the end of the t=0 study visit (Phase 1). Dosing will commence the day after the t=0 study visit. At the end of Phase 1, participants will enter a 'washout' period, when they will cease treatment. After approximately 3 months of washout, participants will cross-over to the other treatment regimen and receive the other interventional product (IP) for the final 6 months of their study participation (Phase 2).
  Other Names: Tamoxifen Citrate
  Arms: Drug: ApoTamox 10mg
Drug: Placebo — placebo comparator
  Arms: Placebo

SUMMARY:
This is a phase 1 / 2, randomized, double-blinded, single cross-over study, with a washout period between treatment regimens, to test the efficacy and safety of tamoxifen therapy to improve motor and respiratory function in males with XLMTM.

DETAILED DESCRIPTION:
Pre-clinical studies in Mtm1 knockout mice (a model of XLMTM) demonstrated prolonged survival, increased motor function (including muscle strength), and improved muscle histopathology with tamoxifen treatment. Based on these data, and the known safety profile of the drug in humans, we hypothesize that tamoxifen treatment will be safe and will improve motor and respiratory function in XLMTM patients. This is a randomized, double-blinded, single crossover clinical trial to test this hypothesis and determine the safety and efficacy of tamoxifen in improving motor and respiratory function in MTM patients. Each subject will serve as his own control during the placebo phase of the study. As treatments for XLMTM are current not available, this study addresses a critical unmet need by testing a therapy that, if effective, may serve as a primary treatment, or in the future as an adjunct to other therapies in development.

ELIGIBILITY:
INCLUSION CRITERIA

1. Male
2. Patients ages 6 months and older may participate.
3. XLMTM resulting from a confirmed mutation in the Myotubularin 1 (MTM1) gene
4. Patients over 18 years of age and parent(s)/legal guardian(s) of patients <18 years of age must provide written informed consent prior to participating in the study and informed assent will be obtained from minors, or at least 7 years of age when required by regulation.
5. Willing and able to comply with all protocol requirements and procedures.

EXCLUSION CRITERIA

1. Other disease which may significantly interfere with the assessment of myotubular myopathy (MTM) and is clearly not related to the disease, at the discretion of the qualified investigator.
2. Has undergone surgery or hospitalization < 3 months before starting TAM4MTM (at t = -3 months), or has surgery scheduled during the 18 months of participation in TAM4MTM, which will impede motor assessments in the opinion of the Investigator.
3. Has a history of thromboembolic events
4. Currently enrolled in a treatment study for XLMTM or receiving treatment with an experimental therapy other than pyridostigmine.
5. Treatment with pyridostigmine for < 6 weeks duration (must be greater than 6 weeks to be included in TAM4MTM).
6. Use of concomitant medication known to inhibit CYP2D6 and/or CYP3A4, including clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, goldenseal and grapefruit, paroxetine, troleandomycin, rifampin, phenobarbital, aminoglutethimide, medroxyprogesterone, amiodarone, haloperidol, indinavir, ritonavir, quinidine, rifampicin, or any selective serotonin reuptake inhibitor (SSRI).
7. Subject has a contraindication to tamoxifen or its ingredients

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Motor Function Measure 32 (MFM32) | Baseline to 15 Months
  Mean change from baseline of Motor Function Measure 32 for subjects aged 4 and older
Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders for subjects aged 2-4 years (CHOP INTEND) | Baseline to 15 months
  Mean change from baseline of Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders for subjects aged 2-4 years
10 meter walk test | Baseline to 15 months
  Mean change from baseline in velocity in 10 meter walk test for ambulant participants

SECONDARY OUTCOMES:
Change in pulmonary function testing scores 1) Forced Expiratory Volume in the first second | Baseline to 15 months
  Mean change from baseline in participants without invasive respiratory support
Change in pulmonary function testing scores 2) Forced Vital Capacity | Baseline to 15 months
  Mean change from baseline in participants without invasive respiratory support
Change in pulmonary function testing scores 3) Peak Cough Flow | Baseline to 15 months
  Mean change from baseline in participants without invasive respiratory support
Change in pulmonary function testing scores 4) Maximum Expiratory Pressure | Baseline to 15 months
  Mean change from baseline in participants without invasive respiratory support
Change in pulmonary function testing scores 5) Maximum Inspiratory Pressure or Sniff Inspiratory Pressure | Baseline to 15 months
  Mean change from baseline in participants without invasive respiratory support
invasive ventilation - time off ventilation | Baseline to 15 months
  Mean change in time off ventilator for participants dependent on invasive respiratory support
Incidence and severity of Adverse Events related to the treatment [ Time Frame: 15 Months ] | Baseline to 15 months
  Incidence of serious adverse events and adverse events throughout the study, as assessed by CTCAE v4.0
micro RNA 133a (miR133a) | Baseline to 15 months
  Assess miR133a as a biomarker of XLMTM

CONTACTS AND LOCATIONS:
Overall Officials: Jame J Dowling, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- United States (2):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - National Institutes of Health, Rockville, Maryland
- Hospital for Sick Children, Toronto, Ontario, Canada
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amburgey K, Tsuchiya E, de Chastonay S, Glueck M, Alverez R, Nguyen CT, Rutkowski A, Hornyak J, Beggs AH, Dowling JJ. A natural history study of X-linked myotubular myopathy. Neurology. 2017 Sep 26;89(13):1355-1364. doi: 10.1212/WNL.0000000000004415. Epub 2017 Aug 25. PMID 28842446
- [Background] Maani N, Sabha N, Rezai K, Ramani A, Groom L, Eltayeb N, Mavandadnejad F, Pang A, Russo G, Brudno M, Haucke V, Dirksen RT, Dowling JJ. Tamoxifen therapy in a murine model of myotubular myopathy. Nat Commun. 2018 Nov 19;9(1):4849. doi: 10.1038/s41467-018-07057-5. PMID 30451841
- [Background] Gayi E, Neff LA, Massana Munoz X, Ismail HM, Sierra M, Mercier T, Decosterd LA, Laporte J, Cowling BS, Dorchies OM, Scapozza L. Tamoxifen prolongs survival and alleviates symptoms in mice with fatal X-linked myotubular myopathy. Nat Commun. 2018 Nov 19;9(1):4848. doi: 10.1038/s41467-018-07058-4. PMID 30451843